CLINICAL TRIAL: NCT00052403
Title: Phase I Study of Monoclonal Antibody Anti-Anb3 Integrin in Patients With Advanced Solid Tumors
Brief Title: Monoclonal Antibody Therapy in Treating Patients With Advanced Solid Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was not successful at recruiting particpants
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Patricia LoRusso, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000258300; WSU-C-2453; NCI-5496
Record Dates: First submitted 2003-01-24; First posted 2003-01-27 (Estimated); Last update posted 2014-01-16 (Estimated); Status verified 2014-01

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — Immunization, Passive; Adjuvants, Immunologic; Antibodies, Monoclonal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: monoclonal antibody anti-anb3 integrin
Procedure: anti-cytokine therapy
Procedure: antiangiogenesis therapy
Procedure: antibody therapy
Procedure: biological response modifier therapy
Procedure: growth factor antagonist therapy
Procedure: monoclonal antibody therapy

SUMMARY:
RATIONALE: Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.

PURPOSE: Phase I trial to study the effectiveness of monoclonal antibody therapy in treating patients who have advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose and recommended phase II dose of monoclonal antibody anti-anb3 integrin in patients with advanced solid tumors.
* Determine the toxic effects of this drug in these patients.
* Determine the pharmacokinetics and pharmacodynamics of this drug in these patients.
* Determine the potential anti-tumor activity of this drug in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive monoclonal antibody anti-anb3 integrin IV over 30 minutes weekly. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of monoclonal antibody anti-anb3 integrin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, additional patients are treated as above at that dose level.

PROJECTED ACCRUAL: A total of 27-33 patients will be accrued for this study within 9-11 months.

ELIGIBILITY:
Inclusion Criteria

DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed solid tumor that is unresponsive to currently available therapies or for which no known effective treatment exists
* Measurable or evaluable disease
* Must have clinical or radiological evidence of disease
* Disease must be accessible to biopsy and imaging studies
* No known brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Eastern Cooperative Oncology Group (ECOG) 0-2

Life expectancy

* At least 3 months

Hematopoietic

* Absolute neutrophil count at least 2,000/mm^3
* Platelet count at least 100,000/mm^3
* No prior bleeding disorder

Hepatic

* Bilirubin no greater than 1.2 mg/dL
* alanine aminotransferase test (ALT) and Aspartate Aminotransferase (AST) no greater than 2.5 times upper limit of normal (ULN)
* Prothrombin time (PT)/ partial thromboplastin time (PTT) no greater than ULN

Renal

* Creatinine less than 1.5 mg/dL OR
* Creatinine clearance at least 60 mL/min

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after study
* Willing to be premedicated for delayed contrast-enhanced MRI
* No prior claustrophobia
* No dementia or altered mental status that would preclude informed consent
* No other uncontrolled concurrent illness
* No ongoing or active infection
* No psychiatric illness or social situations that would preclude study compliance
* No immunodeficiency
* HIV negative
* Must be willing to receive blood products
* No thyroid disease
* Thyroxine and thyroid-stimulating hormone no greater than ULN

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 4 weeks since prior immunotherapy

Exclusion Criteria Chemotherapy

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* Prior taxanes allowed
* No concurrent chemotherapy

Endocrine therapy

* No concurrent hormonal therapy except:
* Concurrent hormonal replacement therapy
* Concurrent medication for maintaining castrate status in patients with progressive hormone refractory prostate cancer

Radiotherapy

* At least 4 weeks since prior radiotherapy and recovered
* No prior radiotherapy to more than 25% of the bone marrow
* No concurrent radiotherapy

Surgery

* More than 4 weeks since prior surgery

Other

* No other concurrent investigational or commercial agents or therapies for the malignancy
* No other concurrent antitumor therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2002-02

CONTACTS AND LOCATIONS:
Overall Officials: Patricia LoRusso, DO, Study Chair — Harper Hospital